CLINICAL TRIAL: NCT05224245
Title: A Study to Evaluate the Feasibility and Safety of the ACURATE Prime™ XL Aortic Valve System in Patients Indicated for TAVI: ACURATE Prime XL Human Feasibility Study
Brief Title: ACURATE Prime XL Human Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: S2458
Record Dates: First submitted 2022-01-04; First posted 2022-02-04 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Aortic Stenosis
Keywords: ACURATE Prime™ XL Aortic Valve System
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Intervention Model Description: The protocol allows for up to 20 patients to be enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm: ACURATE Prime XL Transfemoral Aortic Valve System (Experimental): Subjects who provide written informed consent, meet all eligibility criteria, and are approved by the Case Review Committee (CRC) will be implanted with ACURATE Prime XL Transfemoral Aortic Valve using iSLEEVE, ACURATE Prime XL Delivery System and ACURATE Prime XL Loading kit
  Interventions: Device: ACURATE Prime XL Transfemoral Aortic Valve System

INTERVENTIONS:
Device: ACURATE Prime XL Transfemoral Aortic Valve System — ACURATE Prime™ Transfemoral Aortic Valve system: Support frame made of nitinol, supra-annular processed tri-leaflet porcine pericardial valve and an outer skirt to limit paravalvular regurgitation (manufactured by Boston Scientific Corporation, Marlborough, MA, USA).

SUMMARY:
To evaluate feasibility and safety of the ACURATE Prime™ XL Transfemoral Aortic Valve System for transcatheter aortic valve implantation (TAVI) in subjects with severe native aortic stenosis who are indicated for TAVI.

DETAILED DESCRIPTION:
The ACURATE Prime XL Human Feasibility Study (ACURATE Prime XL HFS) is a prospective, multicenter, open-label, single-arm study designed to evaluate feasibility and safety of the ACURATE Prime XL Transfemoral Aortic Valve System for TAVI in subjects who have severe native aortic stenosis and are indicated for TAVI.

Subjects who provide written informed consent, meet all eligibility criteria, and are approved by the Case Review Committee (CRC) are considered enrolled when an attempt is made to insert the iSLEEVE Introducer into the subject's femoral artery. There will be up to 20 subjects enrolled at up to 6 centers in Australia and Europe.

All subjects implanted with a study valve will be assessed at baseline, peri- and post-procedure, at discharge or 7 days post index procedure (whichever comes first), 30 days, 6 months, and 1 year. Subjects who are enrolled but not implanted with a study valve at the time of the procedure will be followed for safety through 30 days.

ELIGIBILITY:
Inclusion Criteria:

* IC1. Subject has documented severe symptomatic native aortic stenosis defined as follows: aortic valve area (AVA) ≤1.0 cm2 (or AVA index ≤0.6 cm2/m2) AND a mean pressure gradient ≥40 mmHg, OR maximal aortic valve velocity ≥4.0 m/s, OR Doppler velocity index ≤0.25 as measured by echocardiography and/or invasive hemodynamics. Note: In cases of low flow, low gradient aortic stenosis with left ventricular dysfunction (ejection fraction <50%), dobutamine can be used to assess the grade of aortic stenosis (maximum dobutamine dose of 20 mcg/kg/min recommended); the subject may be included in the study if echocardiographic criteria are met with this augmentation.
* IC2. Subject has a documented aortic annulus diameter of ≥26.5 mm and ≤29 mm based on the center's assessment of pre-procedure diagnostic imaging (and confirmed by the Case Review Committee [CRC]).
* IC3. For subjects with symptomatic aortic valve stenosis per IC1 definition above, functional status is NYHA Functional Class ≥ II.
* IC4. Heart team (composition per local standards, but at a minimum must include an experienced cardiac surgeon) agrees that the subject is indicated for TAVI, is likely to benefit from prosthetic valve implantation, and TAVI is appropriate.
* IC5. Subject (or legal representative) understands the study requirements and the treatment procedures and provides written informed consent.
* IC6. Subject, family member, and/or legal representative agree(s) and subject is capable of returning to the study hospital for all required scheduled follow up visits.
* IC7. Subject is expected to be able to take the protocol-required adjunctive pharmacologic therapy.

Exclusion Criteria:

* EC1. Subject has a unicuspid or bicuspid aortic valve.
* EC2. Subject has had an acute myocardial infarction within 30 days prior to the index procedure (defined as Q-wave MI or non-Q-wave MI with total CK elevation ≥ twice normal in the presence of CK MB elevation and/or troponin elevation).
* EC3.Subject has had a cerebrovascular accident or transient ischemic attack clinically confirmed by a neurologist or neuroimaging within the past 6 months prior to study enrollment.
* EC4.Subject has eGFR < 20 mL/min (based on hospital preferred method) but is not on renal replacement therapy.
* EC5. Subject has a pre-existing prosthetic aortic or mitral valve.
* EC6. Subject has severe (4+) aortic, tricuspid, or mitral regurgitation.
* EC7. Subject has moderate or severe mitral stenosis (mitral valve area ≤1.5 cm2 and diastolic pressure half-time ≥150 ms, Stage C or D).
* EC8. Subject has a need for emergency surgery for any reason.
* EC9. Subject has a history of endocarditis within 6 months of index procedure or evidence of an active systemic infection or sepsis.
* EC10. Subject has echocardiographic evidence of new intra-cardiac vegetation or intraventricular or paravalvular thrombus requiring intervention.
* EC11. Subject has platelet count <50,000 cells/mm3 or >700,000 cells/mm3, or white blood cell count <1,000 cells/mm3.
* EC12. Subject has had a gastrointestinal bleed requiring hospitalization or transfusion within the past 3 months or has other clinically significant bleeding diathesis or coagulopathy that would preclude treatment with required antiplatelet regimen or will refuse transfusions.
* EC13. Subject has known hypersensitivity to the following:

  * Contrast agents that cannot be adequately pre-medicated, OR
  * Protocol-required medications (aspirin, all P2Y12 inhibitors, heparin), OR
  * Individual components of the investigational valve and/or delivery system (stainless steel, platinum, iridium, nickel, titanium, or polyethylene terephthalate [PET]).
* EC14. Subject has a life expectancy of less than 12 months due to non-cardiac, comorbid conditions based on the assessment of the investigator at the time of enrollment.
* EC15. Subject has hypertrophic cardiomyopathy.
* EC16. Subject has any therapeutic invasive cardiac or vascular procedure within 30 days prior to the index procedure (except for balloon aortic valvuloplasty, pacemaker implantation, or implantable cardioverter defibrillator implantation, which are allowed).
* EC17. Subject has untreated coronary artery disease, which in the opinion of the treating physician is clinically significant and requires revascularization.
* EC18. Subject has severe left ventricular dysfunction with ejection fraction <20%.
* EC19. Subject is in cardiogenic shock or has hemodynamic instability requiring inotropic support or mechanical support devices.
* EC20. Subject has arterial access that is not acceptable for the study device delivery system as defined in the Instructions For Use.
* EC21. Subject has either of the following:

  * Severe vascular disease that would preclude safe access (e.g., aneurysm with thrombus that cannot be crossed safely; marked tortuosity; significant narrowing of the abdominal aorta; severe unfolding of the thoracic aorta; or thick, protruding, ulcerated atheroma in the aortic arch), OR
  * Severe/eccentric calcification of the aortic annulus that would prevent safe implantation of the TAVI prosthesis.
* EC22. Subject has current problems with substance abuse (e.g., alcohol, etc.) that may interfere with the subject's participation in this study.
* EC23. Subject is participating in another investigational drug or device study that has not reached its primary endpoint or subject intends to participate in another investigational device clinical trial within 12 months after the index procedure.
* EC24. Subject has untreated conduction system disorder (e.g., Type II second degree atrioventricular block) that in the opinion of the treating physician is clinically significant and requires a pacemaker implantation. Enrollment is permissible after permanent pacemaker implantation.
* EC25. Subject has severe incapacitating dementia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2023-05-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with Device Success | Through discharge or 7 days post procedure
  Absence of procedural mortality, AND Correct positioning of a single valve into the proper anatomical location, AND Intended performance of the study device (indexed effective orifice area [iEOA] >0.85 cm2/m2 for BMI <30 kg/m2 and iEOA >0.70 cm2/m2 for BMI ≥30 kg/m2 plus either a mean aortic valve gradient <20 mmHg or a peak velocity <3m/sec, and no moderate or severe prosthetic valve aortic regurgitation) as measured by transthoracic echocardiography (TTE) and assessed by an independent core laboratory.
Number of participants who died or experienced a stroke | Through 30 Days post procedure
  Composite of all-cause mortality and all stroke
  A Clinical Events Committee (CEC), independent group of physician experts will be used to evaluate all reported cases of death and stroke to determine whether they met the specific protocol definition of the event.

OTHER OUTCOMES:
Number of participants who died including all-cause, cardiovascular, and non-cardiovascular death | Participants will be followed for the duration of hospital stay, through 30 days, 6 months, and 1 year
  Adjudicated by an independent Clinical Events Committee (CEC) based on VARC 2 definitions
Number of participants who experienced a Stroke including disabling and non-disabling | Participants will be followed for the duration of hospital stay, through 30 days, 6 months, and 1 year
  Adjudicated by an independent Clinical Events Committee (CEC) based on VARC 2 definitions
Number of participants with Myocardial infarction (MI): periprocedural (≤72 hours post index procedure) and spontaneous (>72 hours post index procedure) | Participants will be followed for the duration of hospital stay, through 30 days, 6 months, and 1 year
  Adjudicated by an independent Clinical Events Committee (CEC) based on VARC 2 definitions
Number of participants with Bleeding: life-threatening (or disabling) and major | Participants will be followed for the duration of hospital stay, through 30 days, 6 months, and 1 year
  Adjudicated by an independent Clinical Events Committee (CEC) based on VARC 2 definitions
Number of participants with Acute kidney injury based on the AKIN System Stage 3 (including renal replacement therapy) or Stage 2 | ≤7 days post index procedure
  Adjudicated by an independent Clinical Events Committee (CEC) based on VARC 2 definitions
Number of participants with Major vascular complication | Participants will be followed for the duration of hospital stay, through 30 days, 6 months, and 1 year
  Adjudicated by an independent Clinical Events Committee (CEC) based on VARC 2 definitions
Number of participants with Repeat procedure for valve-related dysfunction (surgical or interventional therapy) | Participants will be followed for the duration of hospital stay, through 30 days, 6 months, and 1 year
  Adjudicated by an independent Clinical Events Committee (CEC) based on VARC 2 definitions
Number of participants with Hospitalization for valve-related symptoms or worsening congestive heart failure (New York Heart Association [NYHA] class III or IV) | Participants will be followed for the duration of hospital stay, through 30 days, 6 months, and 1 year
  Adjudicated by an independent Clinical Events Committee (CEC) based on VARC 2 definitions
Number of participants with New permanent pacemaker implantation (PPI) resulting from new or worsened conduction disturbances | Participants will be followed for the duration of hospital stay, through 30 days, 6 months, and 1 year
  Adjudicated by an independent Clinical Events Committee (CEC) based on VARC 2 definitions
Number of participants with New onset of atrial fibrillation or atrial flutter | Participants will be followed for the duration of hospital stay, through 30 days, 6 months, and 1 year
  Adjudicated by an independent Clinical Events Committee (CEC) based on VARC 2 definitions
Number of participants with Coronary obstruction: periprocedural | ≤72 hours post index procedure
  Adjudicated by an independent Clinical Events Committee (CEC) based on VARC 2 definitions
Number of participants with Ventricular septal perforation: periprocedural | ≤72 hours post index procedure
  Adjudicated by an independent Clinical Events Committee (CEC) based on VARC 2 definitions
Number of participants with Mitral apparatus damage: periprocedural | ≤72 hours post index procedure
  Adjudicated by an independent Clinical Events Committee (CEC) based on VARC 2 definitions
Number of participants with Cardiac tamponade: periprocedural | ≤72 hours post index procedure
  Adjudicated by an independent Clinical Events Committee (CEC) based on VARC 2 definitions
Number of participants with Valve migration | Participants will be followed for the duration of hospital stay, through 30 days, 6 months, and 1 year
  Adjudicated by an independent Clinical Events Committee (CEC) based on VARC 2 definitions
Number of participants with Valve embolization | Participants will be followed for the duration of hospital stay, through 30 days, 6 months, and 1 year
  Adjudicated by an independent Clinical Events Committee (CEC) based on VARC 2 definitions
Number of participants with Ectopic valve deployment | Participants will be followed for the duration of hospital stay, through 30 days, 6 months, and 1 year
  Adjudicated by an independent Clinical Events Committee (CEC) based on VARC 2 definitions
Number of participants with Transcatheter aortic valve (TAV)-in-TAV deployment | Participants will be followed for the duration of hospital stay, through 30 days, 6 months, and 1 year
  Adjudicated by an independent Clinical Events Committee (CEC) based on VARC 2 definitions
Number of participants with Prosthetic aortic valve thrombosis | Participants will be followed for the duration of hospital stay, through 30 days, 6 months, and 1 year
  Adjudicated by an independent Clinical Events Committee (CEC) based on VARC 2 definitions
Number of participants with Prosthetic aortic valve endocarditis | Participants will be followed for the duration of hospital stay, through 30 days, 6 months, and 1 year
  Adjudicated by an independent Clinical Events Committee (CEC) based on VARC 2 definitions
Number of participants with successful vascular access, delivery and deployment of the study valve, and successful retrieval of the delivery system (site reported assessment) | Participants will be followed for the duration of their procedure, an expected average of 1 day (peri- and post-procedure)
  Device Performance endpoint, as measured by site reported data
Grade of aortic regurgitation/paravalvular leak (PVL) (echocardiographic assessment) | Participants will be followed for the duration of their procedure, an expected average of 1 day (peri- and post-procedure)
  Device Performance endpoint, as assessed by Echocardiographic Core Laboratory
Prosthetic aortic valve performance: Effective Orifice Area (EOA) | Discharge or 7 days post index procedure (whichever comes first), 30 days, 6 months, and 1 year
  Effective Orifice Area (EOA), as measured by transthoracic echocardiography (TTE) and assessed by an independent core laboratory
Prosthetic aortic valve performance: Mean Aortic Gradient | Discharge or 7 days post index procedure (whichever comes first), 30 days, 6 months, and 1 year
  Mean aortic gradient as measured by transthoracic echocardiography (TTE) and assessed by an independent core laboratory
Prosthetic aortic valve performance: Peak Aortic Gradient | Discharge or 7 days post index procedure (whichever comes first), 30 days, 6 months, and 1 year
  Peak Aortic Gradient as measured by transthoracic echocardiography (TTE) and assessed by an independent core laboratory
Prosthetic aortic valve performance: Peak Aortic Velocity | Discharge or 7 days post index procedure (whichever comes first), 30 days, 6 months, and 1 year
  Peak Aortic Velocity as measured by transthoracic echocardiography (TTE) and assessed by an independent core laboratory
Prosthetic aortic valve performance: Grade of Aortic Regurgitation/PVL | Discharge or 7 days post index procedure (whichever comes first), 30 days, 6 months, and 1 year
  Grade of Aortic Regurgitation/PVL as measured by transthoracic echocardiography (TTE) and assessed by an independent core laboratory
Number of participants with a New York Heart Association (NYHA) Functional Status classification of Class I, II, III or IV | Discharge or 7 days post index procedure (whichever comes first), 30 days, 6 months, and 1 year
  Evaluated by New York Heart Association (NYHA) classification
Neurological status: Participant score for National Institutes of Health Stroke Scale (NIHSS) assessment | Discharge or 7 days post index procedure (whichever comes first) and 1 year and when is stroke is suspected
  Evaluated by National Institutes of Health Stroke Scale (NIHSS) - Minimum: 0 (No stroke symptoms); Max: 21-42 (Severe stroke)
Neurological status: Participant score for Modified Rankin Scale (mRS) Assessment | Discharge or 7 days post index procedure (whichever comes first), 30 days, 6 months, and 1 year, and when is stroke is suspected (and 90 days post stroke)
  Evaluated by Modified Rankin Scale (mRS) - min: 0 (The patient has no residual symptoms); max: 6 (The patient has expired)
Neurological status: Number of participants with a confirmed stroke per Neurological physical exam assessment | Participants will be followed for the duration of the trial, through 1 year
  Evaluated per neurological physical exam in all subjects where stroke is suspected

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gooley, MBBS, Principal Investigator — Monash Medical Centre
Locations (3):
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - The Prince Charles Hospital, Brisbane, Queensland
  - Monash Health, Clayton, Victoria

IPD SHARING:
Plan to Share IPD: Undecided
The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy (http://www.bostonscientific.com/en-US/data-sharing-requests.html)

REFERENCES:
- [Derived] Gooley R, Murdoch D, Ng MK, Modolo R, Allocco DJ. First results from the ACURATE Prime XL human feasibility study. Cardiovasc Revasc Med. 2023 Dec;57:1-5. doi: 10.1016/j.carrev.2023.06.028. Epub 2023 Jun 30. PMID 37429793